CLINICAL TRIAL: NCT01834560
Title: Subgenual Cingulate Stimulation in Resistant Depression
Brief Title: SubGenual CG25 Deep Brain Stimulation in Severe Resistant Depression
Acronym: CG25
Status: Completed | Type: Observational
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Other Study IDs: CG25
Record Dates: First submitted 2013-03-21; First posted 2013-04-18 (Estimated); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Depression
Keywords: deep brain stimulation; subgenual cortex (CG25)
MeSH Terms: conditions — Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Despite the availability of several treatments, a number of patients with major depression are refractory to therapeutical approaches and therefore suffer from chronic handicap. For these severe patients, neurosurgical therapies can be envisaged. They aim at interrupting bundles that link the orbitofrontal cortex with striatum and can therefore benefit for the patients.

This study intends to repeat Dr. Lozano's study, published in 2005 in the journal Neuron. In this study, they performed a preliminary evaluation of chronic deep brain stimulation (DBS) of the subgenual cingulate region (Brodmann area 25) to treat refractory depression as an alternative to subcaudate tractotomy. This last technique was employed in Grenoble in the 60s with satisfying results before neurosurgery for psychiatric disorders was abandoned. Since 1992, psychosurgical therapies that respect ethical recommendations have regained interest to treat highly impaired patients. Before the investigators can propose deep brain stimulation of subgenual cingulate brain region as a new therapeutic approach for the investigators patients in Grenoble, the investigators decided to reproduce their clinical evaluation on a group of 6 patients, repeating their methodology faithfully. Therefore nothing was changed to the model used by Drs. Lozano and Mayberg and the investigators took advantage of the investigators own expertise regarding deep brain stimulation and subcaudate tractotomy.

Protocol is strictly identical to the one of Mayberg and Lozano in order to confirm their preliminary results. Cartography of physiological consequences of this procedure will be assessed by measuring cerebral blood flow by PET scan (positron emission tomography). Patients will be monitored and thoroughly assessed during including psychiatric, neurological, neurosurgical, neuropsychological and PET scan exams to measure treatment efficacy and potential adverse reactions. Patients will be followed for two more years to assess medium-term complications. This study will be a first step toward further research including potentially a multicentric clinical trial.

DETAILED DESCRIPTION:
The protocol involves assessment of effects of CG25 (subgenual cingulate area-Brodmann 25) DBS on mood, anxiety, apathy, anhedonia, psychomotor retardation, functional state as well as safety and tolerance by specific psychometric scores.

Moreover the protocol aims at highlighting the neurocircuits modulated by CG25 DBS by means of PET (positron emission tomography) imagery

ELIGIBILITY:
Inclusion criteria:

* Men and women between 30 and 55 years old
* Women at a reproductive age will have to be under successful contraceptive and will undergo a pregnancy test before inclusion
* Patient suffering from major unipolar depression refractory to conventional therapies
* Chronic depression with ongoing depressive episode > 12 months.
* 4 unsuccessful therapies attempted to treat the ongoing episode, including anti-depressant monotherapies, potentialisation of antidepressant treatments, validated structured psychotherapies, electro-convulsive therapy performed accordingly to ANAES ( Agence Nationale d'Accréditation et d'Evaluation en Santé-the French Health Authority) recommendations (at least 6 sessions with bilateral technique and length control of convulsive crisis).
* Ambulatory or hospital care
* Able to speak French, understand study procedures and complete questionnaires.
* Covered by french social health system
* Living in Rhone-Alpes area without plan to move in the next 2 years

Exclusion criteria:

* History of cerebral surgery
* Neurological disorder that can interfere with evaluation of surgical procedure or significant cognitive impairment (Mattis score < 30)
* Psychiatric disorder responsible for comorbidity with the major depressive episode (schizophrenia and other delirium, diagnosed anxiety except generalized anxiety disorder, substance dependency)
* Personality disorder of A and B clusters
* Suicidal ideas at evaluation, intention for auto-destruction, repeated suicidal attempts in the last 3 years with emergency care or hospitalization
* Severe somatic pathology or contraindication to surgery due to heart defibrillator/pacemaker or other implanted device.
* A decrease superior to or equal to 20% in the 17-Hamilton Depression Rating Scale score between inclusion and pre-surgery evaluation
* Drug dependency including alcohol in the last 12 months with history of abuse in the last 6 months, with the exception of nicotine
* Persons protected by the law.

Ages: 30 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: patients suffering from severe depression and referred by the psychiatry department of french University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2007-12; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change from Baseline of the Score at the Hamilton Depression Rating Scale | baseline, at 1 year

SECONDARY OUTCOMES:
neurological examination | monthly during the first 6 mo and every 3 months until the end of the 1st year

OTHER OUTCOMES:
Functional outcome and health status measured by Short Form Health Survey (SF-36) scale | at baseline, at 3 months, 12 months, 24 months
  SF-36 scale assesses both physical and mental health status.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Chabardes, MD, PhD, Principal Investigator — University Hospital, Grenoble
Locations (1):
- Neurosurgery department, Grenoble, France